CLINICAL TRIAL: NCT00773201
Title: Identification of the Genetic Sources of Variability of the Adaptation of the Ventricular Repolarisation at a Pharmacological and Physiological Stimulus in an Apparently Normal Population
Brief Title: Genetic Sources of Variability of the Adaptation of the Ventricular Repolarisation
Acronym: Generepol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P071001
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-06

CONDITIONS: Healthy Volunteers
Keywords: Long QT syndrome; Cardiac repolarisation; Genome-wide association; Electrophysiology; Drugs/adverse effects
MeSH Terms: conditions — Long QT Syndrome | interventions — Sotalol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Healthy subjects
  Interventions: Drug: Sotalol 80 mg

INTERVENTIONS:
Drug: Sotalol 80 mg — healthy subjects will receive an unique dose of Sotalol and will have an effort test on ergonomic bicycle, an auditive stimulation and a taking of DNA

SUMMARY:
The main objective is to research for genetic factors involved in the extreme modifications of the QT interval of the electrocardiogram in answer to a pharmacological stimulation (sotalol) and physiological stimulation in the apparently normal general population.

The phenotypic characterization, based on the ventricular repolarisation dynamics will be used aiming at term of the predictive genetic factors of the acquired long QT syndrome

DETAILED DESCRIPTION:
Study of 1000 apparently healthy subjects which will receive an unique dose of Sotalol and will have an effort test on ergonomic bicycle, an auditive stimulation and a taking of DNA.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Age between 18 and 60 years
* European or North African Origin
* Body mass index between 19 and 29 kg / m ²
* Obtaining informed and written consent

Exclusion Criteria:

* Asthma
* Heart rate < 50 bpm
* Systolic blood pressure < 100 mm Hg
* Atrioventricular block
* Known chronic illness with chronic treatment
* Raynaud phenomenon
* QT prolonging drug
* Family or personal history of the congenital long QT syndrome
* QT/QTc Fridericia (QTcf) > 450 ms
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 997 (Actual)
Dates: Start 2008-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The elongation of the corrected interval QT duration 3 hours after the unique oral taking of an 80 mg dose of Sotalol. | 3 hours after the taking of Sotalol

SECONDARY OUTCOMES:
Constitute a biological base and a phenotypic base of resources which will allow to define answer phenotypes to the implemented dynamic tests | At the inclusion visit
Look for associations between these phenotypes of electrocardiographically answer and mutations or polymorphisms. | At the inclusion visit

CONTACTS AND LOCATIONS:
Overall Officials: Beny Charbit, MD, Principal Investigator — Hôpital Saint Antoine, Assistance Publique - Hopitaux de Paris
Locations (1):
- Centre d'investigation clinique; Hôpital Saint Antoine, Paris, France

REFERENCES:
- [Derived] Salem JE, Germain M, Hulot JS, Voiriot P, Lebourgeois B, Waldura J, Tregouet DA, Charbit B, Funck-Brentano C. GENomE wide analysis of sotalol-induced IKr inhibition during ventricular REPOLarization, "GENEREPOL study": Lack of common variants with large effect sizes. PLoS One. 2017 Aug 11;12(8):e0181875. doi: 10.1371/journal.pone.0181875. eCollection 2017. PMID 28800628